CLINICAL TRIAL: NCT06060704
Title: A Prospective, Open, Single-center, Single-arm Study to Explore Envafolimab Combined With Trifluridine/Tipiracil and Bevacizumab in the Treatment of mCRC Patients Who Were Refractory to Second-line and Above Standard Therapy.
Brief Title: Envafolimab Combined With Trifluridine/Tipiracil and Bevacizumab in the Treatment of Refractory mCRC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 09
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — envafolimab; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Envafolimab Combined With Trifluridine/Tipiracil and Bevacizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- triplet combination therapy (Experimental): Envafolimab Combined With Trifluridine/Tipiracil and Bevacizumab
  Interventions: Drug: Envafolimab; Drug: Trifluridine/Tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Envafolimab — 150mg Qw, delivered as a single 1.5ml subcutaneous injection in under 30s , every 4 weeks for one cycle(Q4w).
Drug: Trifluridine/Tipiracil — 35 mg/m2 (maximum single dose of 80 mg), po, on days 1-5 and 8-12 of each treatment cycle, twice daily for 28 days, within 1 hour after breakfast or dinner take medicine.
  Other Names: TAS-102; FTD/TPI
Drug: Bevacizumab — ivgtt, 5mg/kg, d1, d15, every 4 weeks for one cycle (Q4w). The subjects will receive Trifluridine/Tipiracil plus Bevacizumab and Envafolimab until disease progression, intolerable toxicity, initiation of other anti-tumor therapy, death, withdrawal of informed consent, or loss of follow-up.

SUMMARY:
The goal of this single-arm study is to evaluate the efficacy and safety of Envafolimab combined with Trifluridine/Tipiracil and Bevacizumab in the treatment of metastatic colorectal cancer patients who are refractory or intolerant to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient able and willing to provide written informed consent and to comply with the study protocol and follow-up inspection.
* Histologically or cytologically documented diagnosis of metastatic colorectal cancer refractory to second-line and above standard treatment; presence of at least one measurable lesions which should be measured on CT or MRI following RECIST 1.1 criteria.
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2.
* Life expectancy of at least 3 months.
* Patient had no serious hematologic,hepatic, or renal abnormalities, and the results within a week were consistent with the following laboratory tests:

  1. Hematological Parameters: Neutrophil count ≥1.5×109/L;Platelets ≥80×109/L;Hemoglobin≥90g/L.
  2. Hepatic Function Parameters: AST and ALT ≤2.5×upper limit of normal（≤5×ULN if liver metastasis present）; Bilirubin ≤2.5 ×upper limit of normal.
  3. Renal Function Parameters: Cr ≤ 1.5×upper limit of normal.
  4. Coagulation Function Parameters: International Normalized Ratio (INR)≤1.5 or prothrombin time (PT)≤1.5×ULN or activated partial prothrombin time (APTT)≤1.5×ULN.
  5. Urinary protein≤1+, 24-hour urinary protein quantity ≤1.0g.

Exclusion Criteria:

* Symptomatic or known central nervous system metastases (head CT or MRI is not required to rule out brain metastases). For patients with suspected neurological metastasis, head CT or MRI should be performed within 28 days before enrollment to rule out neurological metastasis.
* The target lesion was treated locally within 3 months.
* There are neurological or psychiatric abnormalities that affect cognitive ability.
* Subjects with hypertension not well controlled by single antihypertensive medication (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg); Patients with history of unstable angina pectoris; Patients with newly diagnosed angina pectoris or myocardial infarction within 3 months prior to screening; Arrhythmias (including QTcF: ≥450 ms in men and ≥470 ms inwomen) require long-term use of antiarrhythmic drugs and New York Heart Association grade ≥II cardiac insufficiency.
* Prior or combined history of other malignancies, with the exception of cured basal cell carcinoma of the skin,carcinoma in situ of the cervix, and other early tumors that are expected to be free of recurrence within six months after radical treatment.
* Patients currently receiving or having received anticancer therapies within 4 weeks prior to the enrollment.
* For female subjects: should be surgically sterilized, postmenopausal, or consent to use a medically approved contraceptive during the study treatment and for 6 months after the end of the study treatment period; Serum or urine pregnancy tests must be negative within 7days prior to study enrollment and must be non-lactating. Male subjects: Patients who should be surgically sterilized or who have consented to use a medically approved contraceptive method during the study treatment period and for 6 months after the end of the study treatment period.
* There are multiple factors that affect oral medications (such as inability to swallow,chronic diarrhea, and intestinal obstruction).
* Patients with active bleeding, long-term unhealed wounds, and any surgical procedures within 2 months.
* Any arteriovenous thrombosis event occurred within 6 months, including cerebrovascular accident, deep vein thrombosis (deep vein thrombosis caused by the installation of a deep vein catheter in the previous chemotherapy, except for those who were judged to have recovered by the investigator), and pulmonary embolism.
* Severe chest and abdominal fluid, requiring clinical intervention.
* Have thyroid dysfunction that cannot be maintained within the normal range despite medication.
* History of immune deficiency or organ transplantation.
* There were other concomitant diseases that the investigators determined to seriously endanger the patient's safety or interfere with the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
ORR（Objective response rate） | Approximately 12 months
  Objective Response Rate defined as the proportion of patients with objective evidence of complete response (CR) or partial response (PR) according to RECIST version 1.1 criteria and using investigator's tumor assessment.

SECONDARY OUTCOMES:
OS (Overall Survival) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of first treatment and the date of death due to any cause.
PFS (Progression-free survival) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the randomization and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.
DCR (Disease control rate) | Approximately 12 months
  Disease control rate defined as the proportion of patients with objective evidence of CR or PR or stable disease (SD) according to RECIST version 1.1 criteria and using investigator's tumor assessment.
Quality of life: EORTC QLQ-C30 | Approximately 12 months
  Assess patients health and activities using the European Organization for Research and Treatment of Cancer Core Quality of Life (EORTC QLQ-C30) module.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Gu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No